CLINICAL TRIAL: NCT03387345
Title: β-glucan Rich Barley and Rice Mixes and Post-prandial Glycemia - a Dose Response Study
Brief Title: Barley and Rice Mixture Effects on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Ardent Mills, LLC (Unknown)
Responsible Party: Principal Investigator, Corrie Whisner, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005413
Record Dates: First submitted 2017-12-19; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Blood Glucose; Dietary Fiber; Hunger
Keywords: glucose; dietary fiber; glycemia; whole grain

STUDY DESIGN:
Intervention Model Description: Otherwise healthy male and female adults
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- bread-50/50-steelcut-80/20-flake-rice (Experimental): 25 g of available carbohydrate was delivered to participants via (1) white bread, followed by (2) 50/50 rice-barley mix, followed by (3) 100% steel cut barley, followed by (4) 80/20 rice-barley mix, followed by (5) 100% barley flakes, followed by (6) 100% rice
  Interventions: Other: 100% steel cut barley; Other: 100% barley flakes; Other: 50/50 rice-barley mix; Other: 80/20 rice-barley mix; Other: 100% rice; Other: white bread
- 50/50-steelcut-80/20-flake-rice-bread (Experimental): 25 g of available carbohydrate was delivered to participants via (1) 50/50 rice-barley mix, followed by (2) 100% steel cut barley, followed by (3) 80/20 rice-barley mix, followed by (4) 100% barley flakes, followed by (5) 100% rice, followed by (6) white bread
  Interventions: Other: 100% steel cut barley; Other: 100% barley flakes; Other: 50/50 rice-barley mix; Other: 80/20 rice-barley mix; Other: 100% rice; Other: white bread
- steelcut-80/20-flake-rice-bread-50/50 (Experimental): 25 g of available carbohydrate was delivered to participants via (1) 100% steel cut barley, followed by (2) 80/20 rice-barley mix, followed by (3) 100% barley flakes, followed by (4) 100% rice, followed by (5) white bread, followed by (6) 50/50 rice-barley mix
  Interventions: Other: 100% steel cut barley; Other: 100% barley flakes; Other: 50/50 rice-barley mix; Other: 80/20 rice-barley mix; Other: 100% rice; Other: white bread
- 80/20-flake-rice-bread-50/50-steelcut (Experimental): 25 g of available carbohydrate was delivered to participants via (1) 80/20 rice-barley mix, followed by (2) 100% barley flakes, followed by (3) 100% rice, followed by (4) white bread, followed by (5) 50/50 rice-barley mix, followed by (6) 100% steel cut barley
  Interventions: Other: 100% steel cut barley; Other: 100% barley flakes; Other: 50/50 rice-barley mix; Other: 80/20 rice-barley mix; Other: 100% rice; Other: white bread
- flake-rice-bread-50/50-steelcut-80/20 (Experimental): 25 g of available carbohydrate was delivered to participants via (1) 100% barley flakes, followed by (2) 100% rice, followed by (3) white bread, followed by (4) 50/50 rice-barley mix, followed by (5) 100% steel cut barley, followed by (6) 80/20 rice-barley mix
  Interventions: Other: 100% steel cut barley; Other: 100% barley flakes; Other: 50/50 rice-barley mix; Other: 80/20 rice-barley mix; Other: 100% rice; Other: white bread
- rice-bread-50/50-steelcut-80/20-flake (Experimental): 25 g of available carbohydrate was delivered to participants via (1) 100% rice, followed by (2) white bread, followed by (3) 50/50 rice-barley mix, followed by (4) 100% steel cut barley, followed by (5) 80/20 rice-barley mix, followed by (6) 100% barley flakes
  Interventions: Other: 100% steel cut barley; Other: 100% barley flakes; Other: 50/50 rice-barley mix; Other: 80/20 rice-barley mix; Other: 100% rice; Other: white bread

INTERVENTIONS:
Other: 100% steel cut barley — 25 g of available carbohydrate was delivered to participants via steel cut Sustagrain barley (Ardent Mills, LLC).
Other: 100% barley flakes — 25 g of available carbohydrate was delivered to participants via Sustagrain barley flakes (Ardent Mills, LLC).
Other: 50/50 rice-barley mix — 25 g of available carbohydrate was delivered to participants via a 50/50 mixture (by weight) of Goya medium grain white rice and steel cut Sustagrain barley (Ardent Mills, LLC).
Other: 80/20 rice-barley mix — 25 g of available carbohydrate was delivered to participants via a 80/20 mixture (by weight) of Goya medium grain white rice and steel cut Sustagrain barley (Ardent Mills, LLC).
Other: 100% rice — 25 g of available carbohydrate was delivered to participants via Goya medium grain white rice
Other: white bread — 25 g of available carbohydrate was delivered to participants via Sara Lee Classic White Bread (Bimbo Bakeries USA, Inc.)

SUMMARY:
The purpose of this research was to investigate 5 different formulations of whole grain barley and refined white rice against a control of white bread on post-prandial glycemic response, as well as self-reported hunger/satiety in a randomized cross-over trial.

DETAILED DESCRIPTION:
Beta-glucan-rich barley has been shown to improve glycemic response, reduce hunger and increase satiety. Nutrient-dense grain mixtures that include a new cultivar of barley (Sustagrain, Ardent Mills, LLC) with exceptionally high dietary fiber content may help individuals meet their dietary fiber needs while minimizing the rapid increase in blood glucose following the consumption of a refined grain product. The primary objective of this study was to compare the effects of five different test meals containing varying amounts of whole-grain barley and refined white rice to white bread on post-prandial blood glucose concentrations. A secondary aim was to evaluate changes in self-reported hunger and satiety following the consumption of each treatment. This study was a single-site, blinded, randomized crossover trial among 24 healthy adults. Each participant consumed the following treatments: 100% Sustagrain barley flakes, 100% Sustagrain steel cut barley , an 80/20 rice-steel cut Sustagrain barley mix, a 50/50 rice-steel cut Sustagrain barley mix, 100% rice, and white bread.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, English speaking adults;
* BMI between 18 and 30 kg/m2

Exclusion Criteria:

* History of GI malabsorption diseases, food allergy or intolerance to gluten;
* Prediabetes, and/or diabetes, and/or treatment with diabetic medications for any reason;
* Hypertension, hypothyroidism and other chronic disease that affects nutrient metabolism;
* Any women pregnant or lactating, or expecting to become pregnant during the study;
* Individuals with a history of bleeding disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-18 (Actual)

PRIMARY OUTCOMES:
Post-prandial glycemia | 0 min, 15 min, 30 min, 45min , 60 min, 90 min, 120 min
  Incremental area under the curve(iAUC) for plasma glucose concentrations were measured at 0, 15, 30, 45, 60, 90 and 120 min using the trapezoidal method to evaluate the glycemic response to each grain treatment.

SECONDARY OUTCOMES:
Self-reported hunger | 0 min, 15 min, 30 min, 60 min, 90 min, 120 min
  Visual analog scales were used to evaluate self-reported feelings of hunger using the question "How hungry do you feel?" The scale consisted of a 100-millimeter line with anchors "I am not hungry at all" and "I have never been more hungry" at 0 and 100 millimeters, respectively. Lower numbers represent low feelings of hunger while larger values are characteristic of greater hunger. Hunger was assessed at 0, 15, 30, 60, 90 and 120 minutes to evaluate changes across time for each grain treatment.
Self-reported satiety | 0 min, 15 min, 30 min, 60 min, 90 min, 120 min
  Visual analog scales were used to evaluate self-reported feelings of satiety using the question "How satisfied do you feel?" The scale consisted of a 100-millimeter line with anchors "I am completely empty" and "I cannot eat another bite" at 0 and 100 millimeters, respectively. Lower numbers represent low feelings of satiety while larger values are characteristic of greater satiety. Satiety was assessed at 0, 15, 30, 60, 90 and 120 minutes to evaluate changes across time for each grain treatment.
Self-reported fullness | 0 min, 15 min, 30 min, 60 min, 90 min, 120 min
  Visual analog scales were used to evaluate self-reported feelings of fullness using the question "How full do you feel?" The scale consisted of a 100-millimeter line with anchors "Not at all full" and "Totally full" at 0 and 100 millimeters, respectively. Lower numbers represent low feelings of fullness while larger values are characteristic of greater fullness. Fullness was assessed at 0, 15, 30, 60, 90 and 120 minutes to evaluate changes across time for each grain treatment.
Self-reported prospective food consumption | 0 min, 15 min, 30 min, 60 min, 90 min, 120 min
  Visual analog scales were used to evaluate self-reported feelings toward prospective food consumption using the question "How much do you think you can eat?" The scale consisted of a 100-millimeter line with anchors "Nothing at all" and "A lot" at 0 and 100 millimeters, respectively. Lower numbers represent low ability to eat while larger values are characteristic of greater ability to eat. Prospective food consumption was assessed at 0, 15, 30, 60, 90 and 120 minutes to evaluate changes across time for each grain treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Corrie M Whisner, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No